CLINICAL TRIAL: NCT01823250
Title: Culturally Informed Family Based Treatment of Adolescents: A Randomized Trial
Acronym: CIFFTA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Daniel A. Santisteban, Ph.D., Clinical Psychologist/Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20100055; R01DA027920-01 (NIH)
Record Dates: First submitted 2012-06-11; First posted 2013-04-04 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Substance Use Disorders; Risk Behavior; Psychiatric Disorders; Family Dysfunction
Keywords: Hispanic; adolescent; drug abuse treatment; evidence-based; family therapy; adaptive family treatment; Culturally Informed Family-Based Treatment for Adolescents
MeSH Terms: conditions — Substance-Related Disorders; Risk-Taking; Mental Disorders | interventions — Psychotherapy, Group

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CIFFTA (Experimental): Culturally Informed and Flexible Family-Based Treatment for Adolescents (CIFFTA)involves four months of intervention. Adolescents and families receive one family therapy session per week and an additional session which is either a psycho-educational session for the adolescent and/or parents, or an individual therapy session with the adolescent. There is a total of 2 sessions per week.
  Interventions: Behavioral: Family Therapy based on Structural Family Therapy; Behavioral: Psychoeducational Sessions; Behavioral: Individual Adolescent Therapy Sessions
- Traditional Family Therapy (TFT) (Active Comparator): The Traditional Family Therapy condition consists of once per week family therapy based on Structural Family Theory and a didactic group intervention once per week in which HIV/STI risk is discussed.
  Interventions: Behavioral: Family Therapy based on Structural Family Therapy; Behavioral: Group Therapy

INTERVENTIONS:
Behavioral: Family Therapy based on Structural Family Therapy — Once per week family therapy based on Structural Family Therapy. Sees to improve parenting practices, communication, and problem solving skills. It also seeks to increase the attachment/bond between parents and adolescents.
Behavioral: Group Therapy — Group Therapy is provided once per week and is designed to share information on HIV and STI risk and protection. There are typically 8-10 adolescents in a group.
  Arms: Traditional Family Therapy (TFT)
Behavioral: Psychoeducational Sessions — Psycho-educational sessions are used to provide didactic in formation to parents alone, adolescents alone, or both together. Content may focus on parenting, drug use risks, depression, HIV/STI risk or other major issues that adolescents and families confront. There are also modules that focus on culture-related stressors and processes that can be provided to families for whom this is a prominent issue.
  Arms: CIFFTA
Behavioral: Individual Adolescent Therapy Sessions — Individual sessions with the adolescent focus on Motivational Interviewing, coaching for family sessions, and monitoring of unhealthy behaviors.
  Arms: CIFFTA

SUMMARY:
This Stage II randomized trial tests Culturally Informed & Flexible Family Based Treatment for Adolescents (CIFFTA) developed as part of a Stage I treatment development effort and yielding promising preliminary findings. Drug use rates are highest among Hispanic middle school youth and to date no treatments have met criteria for "Well Established" in the treatment of substance abuse in Hispanic adolescents. Further treatment for Hispanic youth and families is complicated by the fact that these families often differ from mainstream populations in culture-related values, beliefs and behaviors that can directly impact engagement, retention, and efficacy/effectiveness of drug treatment. Our efforts to develop a more powerful treatment capable of addressing these issues began with a Stage 1 study that led to the development of a multi-component treatment that includes a flexible manual that allows treatment tailoring to the unique characteristics of individual families. CIFFTA integrates innovative culturally-based, individually-based, and family-based components to: 1) reduce maladaptive family processes (e.g., poor parenting practices, family conflict) and increase family protective factors (e.g., strong parent-child attachment), 2) teach adolescents skills to effectively manage interpersonal conflicts and stressors and to increase motivation to change, 3) deliver psycho-educational and culturally congruent material (e.g., modules on immigration stressors) to youth and parents both separately and together, and 4) deliver the intervention using a flexible treatment manual that allows the clinician to tailor the treatment (e.g., by selecting the most relevant psycho-educational modules and themes) to the unique characteristics and needs of the Hispanic family.

This Stage II randomized trial randomizes 220 Hispanic adolescents ages 14-17 who meet DSM-IV criteria for Substance Abuse to a 4-month treatment of either CIFFTA or Traditional Family Therapy. The study tests CIFFTA's efficacy in impacting drug use, risky sexual behavior, and other severe behavior problems, and hypothesized mechanisms of change, in a larger and more rigorous Stage II trial. Assessments occur at baseline, 4 months post baseline (end of treatment), 10 months post baseline and 16 months post baseline. Should this line of research continue to be successful, it has the potential to contribute to the field a highly innovative and efficacious treatment for Hispanic drug abusing adolescents, a better understanding of mechanisms of treatment efficacy, and also a framework for future flexible and tailored treatments that can be used to better address the unique needs of other special populations.

DETAILED DESCRIPTION:
This Stage II randomized trial provides a more rigorous test for Culturally Informed & Flexible Family Based Treatment for Adolescents (CIFFTA) which was developed as part of a Stage I treatment development effort and yielded promising preliminary findings. Drug use rates are highest among Hispanic middle school youth and to date no treatments have met criteria for "Well Established" in the treatment of substance abuse in Hispanic adolescents. Further treatment for Hispanic youth and families is complicated by the fact that these families often differ from mainstream populations in culture-related values, beliefs and behaviors that can directly impact engagement, retention, and efficacy/effectiveness of drug treatment. Our efforts to develop a more powerful treatment began with a Stage 1 study that led to the development of a multi-component treatment that includes a flexible manual that allows treatment tailoring to the unique characteristics of individual families. The current Stage II trial randomizes 220 Hispanic adolescents ages 14-17 who meet DSM-IV criteria for Substance Abuse to a 4-month treatment of either CIFFTA or Traditional Family Therapy. The study tests CIFFTA's efficacy in impacting drug use, risky sexual behavior, and other severe behavior problems, and hypothesized mechanisms of change. Should this line of research continue to be successful, it has the potential to contribute to the field a highly innovative and efficacious treatment for Hispanic drug abusing adolescents, a better understanding of mechanisms of treatment efficacy, and also a framework for future flexible and tailored treatments that can be used to better address the unique needs of other special populations.

Design and Methods: The study is divided into three phases. The first phase (months 1- 5) prior to the initiation of the randomized trial focused on: 1) clarifying manual sections and finalizing all assessment measures, 2) hiring and training therapists and assessors, and 3) setting up the web-based data collection system. The second phase (months 6-47) includes the implementation of the randomized trial and the delivery of all clinical treatments. Beginning in month 6 we began to recruit 220 Hispanic adolescents (14-17 years of age) who meet DSM-IV criteria for Substance Abuse or Dependency. Following screening, consent and assessment, the adolescents and their families will be randomly assigned to either the (1) Culturally Informed and Flexible Family-Based Treatment for Adolescents (CIFFTA) or to our Traditional Family Therapy (TFT). The two conditions will be tested as a four month intervention with two sessions per week. The participation of adolescents and families in clinical services will end at approximately month 48 of the grant. The third phase (months 48-60) will focus on the completion of all follow-up assessments, data cleaning and logic checks, data base locks, and the analysis, interpretation and reporting of findings. Assessments will be conducted at baseline, termination (4 months), 6 month follow-up (10 months post baseline), and 12 month follow-up (16 months post baseline). Data from urine analyses, self-reports of therapeutic alliance and data on service utilization outside of the program, will also be collected throughout the entire course of therapy and service utilization will continue during periods between follow-up assessments. Longitudinal data analysis (growth curve modeling) will be used to test study hypotheses. More detail on the details of the randomized trial procedures is provided below.

Randomized Study Design. This is a randomized clinical trial in which 220 14-17 year old Hispanic adolescents meeting DSM-IV criteria for Substance Abuse, and their families will be assessed at baseline, randomized to one of two outpatient conditions (CIFFTA or TFT) in which they will receive treatment twice weekly for four months, and assessed again following termination, 6 months following termination (T3) and 12 months following termination (T4). Randomization will be stratified by gender, number of comorbid psychiatric disorders, whether or not they were mandated to treatment, and whether or not they are taking medication upon entry into the program.

Inclusion of Family members in the study. The target adolescents and parents/guardians are asked to participate in all assessments and in treatment. All other family members living in the household of the target adolescent will be invited to participate in the family treatment but not in assessments. Our previous projects have been very successful at identifying and engaging family members into treatment as well as in retaining them throughout the course of the treatment. In our Stage I project we were successful at engaging family members into treatment as indicated by the fact that we had an average of three family members per participant household participating in the family intervention component.

Participant Recruitment Plan: We have a strong partnership with the Miami Behavioral Health Center which runs the Miami-Dade County Juvenile Addiction Receiving Facility in which all youth meet DSM-IV criteria for drug abuse and for which approximately 80% of the youth are Hispanic. Our previous research projects received many referrals from the JARF and this is bound to increase now that it is located at our partner agency. In our currently NCMHD prevention study with 11-14 year old Hispanic youth and their parents we have been very successful at recruiting from community clinics, middle school counselors, trust counselors and directly from the community. One highly successful strategy was to conduct an interview about the research program on Spanish language television. This strategy used at the initiation of randomization produced a large wave of interested families to the project and facilitated the prompt filling of all slots. Similar interventions on Spanish radio have been equally effective. These strategies will be utilized if participation rates are low.

Screening and Assessment Procedures. Study personnel are trained to identify substance abusing youth and families and to explain the research study in detail. Those interested will be asked to sign an informed consent that allows the screening of inclusion/exclusion criteria. Those individual who meet screening criteria go on to the baseline part of the assessment. Participants that do not meet criteria will receive another set of placement referrals. Participants will be randomized immediately after baseline testing and will be given the name of the therapist that will be contacting them to schedule the first therapy session. All participants will be assessed 4 months after baseline (post-treatment - T2), 10 months after baseline (Follow-up 1 or T3) and 16 months after baseline (Follow-up 2 - T4). All assessments will be administered by highly trained and competent Master's level research assistants who are bilingual in English and Spanish. Our assessors have worked on multiple projects using the same types of self-report and interview measures proposed in this study. All measures and consents will be available in both English Spanish to ensure that primarily Spanish-speaking adolescents or parents are not excluded.

Each assessment interview lasts approximately 3 hours and consists of three parts: an individual interview with the adolescent, an individual interview with each parent, and a family interview session. To ensure participation at the T2-T4 assessments, families will be paid $40 for T2 and $75 for T3 and $100 for T4, for completed assessments. The fees may be slightly higher than other projects that work only with individual participants because our assessments include multiple family members (typically an adolescent and two caregivers). The fee is meant to compensate 3 participants X approximately 3 hours each or 9 total hours of assessment time per time-point. All assessment data are entered directly into a web-based Velos system.

Therapist Supervision and Adherence Monitoring. Separate weekly clinical meetings are held for the CIFFTA and TFT condition therapists. Each therapist will receive formal supervision in these meetings, in addition to consults as needed. Recorded sessions will be reviewed, the clinical complexity of cases will be discussed, and good manual implementation will be emphasized. These meetings help to ensure that manualized interventions are delivered competently. The independent adherence rater will randomly select 20% of the sessions from each condition at different treatment phases (early, mid, and late) for adherence ratings. These rating will document the adequacy with which treatment sessions follow specific manual interventions and treatment strategies. Ratings that fall below adequacy on any dimension/component will trigger increased supervision focus for that dimension and if necessary, re-training. Adherence raters will be trained using the established adherence checklists for the two study conditions which have been developed and used successfully in previous studies. The condition supervisors will be held as the gold-standard for inter-rater reliability on adherence ratings and raters will be trained to achieve an intra-class correlation coefficient of .70 or higher, and at least 80% agreement across items. Inter-rater reliability will be checked regularly to avoid drift.

Prevention of Dropouts from the study. To ensure retaining as much of the sample as possible, each participant will have contact with the same assessment specialist over the entire course of the study. Additional procedures that we have established to retain Ss in the study, and ensure follow-up assessments, include: 1) conducting assessments at convenient locations for the families including their homes when necessary, 2) paying families for their participation in assessments, 3) conducting additional service utilization phone interviews at points between the formal assessment points that is, at 6, 8, 12, and 14 months post-baseline, 4) updating all contact information at regular intervals, and 5) obtaining the names of three contact persons who are close to family members and who may be contacted by the Assessment Specialist in the event that the family is unreachable at the assessment time-points (this is included in the consent form).

Treatment Conditions:

Traditional Family Therapy (TFT). The TFT condition is intended to control for many of the factors present in CIFFTA except for the systematic integration of individual level work and psycho-educational modules within a flexible treatment package. This is the same control intervention that was used in the Stage I study with one exception. In that Stage I study we tested the "add on" effect of the new treatment components and flexibility, to investigate whether such additions would lead to a significant boost in treatment effects. The dosages of the two interventions were not equal. To provide a more rigorous test of the intervention by having equivalent dosages in the two conditions, we have added to the TFT intervention used in the Stage I study, an additional hour per week. The additional weekly hour consists of drug education and risky sexual behavior/STI/HIV information delivered to the youth in a group format. This additional hour per week per client of intervention was selected after consultation with the director of one of the largest local community treatment agencies that uses this approach as a standard of care. The Traditional Family Therapy (TFT) condition intervention is rooted in the Structural Family Therapy work of Salvador Minuchin. TFT is designed to: 1) target behavior problems and substance abuse; and 2) target youth who were unwilling to seek treatment on their own. The typical length of intervention for TFT is 4 months of weekly family sessions. An important assumption underlying this and other family-oriented models is that the family therapist can spend only a limited number of hours with participants, but by changing the family system (parents, extended family, non-blood kin), the family context becomes a force that will positively influence the youth on an around the clock basis.

Culturally Informed and Flexible Family-Based Treatment for Adolescents (CIFFTA). The CIFFTA treatment model has three major components - Family Therapy, Individual Therapy, and Psycho-educational Modules - delivered over 16 weeks in a two session (60 minutes each) per week format. One session will typically be a family session which may include Family Therapy or Psycho-educational modules designed for the family or parents alone. The other session is typically with the adolescent alone, which may include individual treatment or Psycho-educational modules designed for the adolescent. CIFFTA is a flexible manual because it allows for the selection of psycho-educational modules that address specific family and adolescent clinical and cultural issues that are central to that lives of that family. CIFFTA is an outpatient treatment. Home visits although infrequent, may be critically important at times when a key member has disengaged from therapy and must be re-engaged. Visits to schools, courts, and other important institutions in the adolescent's ecology are also allowed as needed (usually a maximum of 2-3 such visits per family).

Individual characteristics that are targeted for modification by CIFFTA include: a) impulsive involvement in unhealthy behaviors such as drug use, risky sexual behavior, and criminal activity, and b) co-occurring psychiatric disorders.

Individual level factors that support healthy development and are promoted by revised CIFFTA will be: 1) increased motivation to work toward healthy development, 2) life skills acquisition, 3) goal setting, 4) knowledge of short and long term drug effects and HIV risk, and 4) improved decision making.

Family characteristics that will be targeted for modification by CIFFTA include: a) maladaptive responses to immigration and acculturation processes and stresses, b) parental neglect, c) verbal or physical violence, and d) interactions that reward/reinforce maladaptive behaviors (i.e., coercive processes).

Family level factors that support healthy development and are promoted by revised CIFFTA will be improvements in: 1) parenting practices, 2) parent-adolescent attachment, 3) parental guidance and leadership, 4) stability of home environment, 5) directness and clarity of communication, and 6) positive/supportive family interactions.

Individual and family level targets of change must be specifically able to address the ecological factors as well. For example, parenting practices may be improved to better monitor the adolescent's peers; parental leadership and guidance may focus on taking a more active role in advocacy in schools; and adolescent skills may become important in better addressing peer pressure in the peer context.

CIFFTA Thematic Psycho-Educational Modules Component The thematic modules component of CIFFTA provides parents and adolescents with focused information/educational sessions on specific areas that are relevant to the family. Content and process are both emphasized during the session, however content is more heavily emphasized in modules while process work (e.g., shaping better communication, deepening their understanding of each other, processing past traumas) is more heavily emphasized in family sessions.

ELIGIBILITY:
Inclusion Criteria:

* The adolescent has a substance abuse disorder,
* The adolescent is 14 to 17 years old, and
* The adolescent is living with at least one family member of an older generation born in a Spanish-speaking country such as a parent or grandparent

Exclusion Criteria:

* History of any of the following DSM IV diagnoses:
* Developmental Disorders
* Elective Mutism
* Organic Mental Disorders (except Psychoactive Substance-Induced)
* Schizophrenia
* Delusional (Paranoid) Disorder
* Psychotic Disorder
* Bipolar Affective Disorder

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 190 (Actual)
Dates: Start 2011-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in Adolescent Drug Use | At baseline, twice per month during the 4 month treatment phase (collection weeks randomly assigned), and 4, 10, and 16 months post baseline.
  Drug use will be assessed using the Time-Line Follow-Back Drug Use Recording Method (TLFB) and a Urine Drug Screen kit. The latter is a self contained testing unit which combines a temperature sensitive collection cup with built in assays for sample adulterants and 9 specific drugs of abuse. The TLFB has been adapted for adolescents and obtains retrospective adolescent reports of daily substance use by using a calendar to stimulate recall. It gathers information on specific substances used, amount of use, social context of use, location of use, and subjective experience of use.

SECONDARY OUTCOMES:
Changes in Service Utilization Interview (SUI) | At baseline and 4, 10, and 16 months post randomization.
  The SUI documents mental health and family services received from 11 types of professionals (e.g. psychologist, psychiatrist) and 15 kinds of groups (e.g. church group, support group), and frequency, reason, and duration of service. Additionally, the SUI captures whether or not any family member has been in contact with law enforcement or the courts (Center for Family Studies, 1995). The SUI (mental health and legal) will be administered to parents at all the formal time-points, and 6, 8, 12 and 14 month post-baseline calls. The SUI takes 15 minutes to complete.
Change in Personal Experiences Inventory (PEI) | At baseline and 4, 10, and 16 months post randomization.
  The PEI is an adolescent self-report measure of involvement with drugs, and degree of psychological and social consequences that takes 10 minutes to complete. Its well-documented psychometric properties are satisfactory (Winters & Henly, 1989).
Change in Risky Sexual Behavior (SRB) | At baseline and 4, 10, and 16 months post randomization.
  Questions ask about the adolescent's number of sexual partners in the past 3 months, frequency of engagement in oral, anal and vaginal intercourse over the past 3 months, and for each occurrence how many times a condom was used, and how many times they were high on alcohol and/or drugs. In our work with Hispanic adolescents, scales for HIV knowledge and intentions showed acceptable internal consistency (alpha) coefficients (.66 to .76).
Change in Behavior Problem Checklist (RBPC) | At baseline and 4, 10, and 16 months post randomization.
  The RBPC (Quay & Peterson, 1987) assesses problem behaviors as reported by parents. Three subscales (50 items) will be used in this study: Conduct Disorder, Socialized Aggression, and Anxiety/Withdrawal. Adolescent problem behaviors are rated (0 = No problem; 1 = mild problem; 2 = severe problem).Psychometric properties with Spanish speaking patients found to be adequate: internal consistency (alpha) coefficients above .89, test-retest reliability coefficients between .49 and .83, and inter-parent reliability between .59 and .87.
Change in Youth Self-Report (YSR) | At baseline and 4, 10, and 16 months post randomization.
  The YSR (Achenbach, 1991) is an adolescent (11-18 years old) self-report instrument that assesses the severity of 119 problem behaviors, and the degree of functioning on three dimensions of Social Competence. Problem behaviors can be scored on the super-ordinate domains of "internalizing" and "externalizing" behaviors, or smaller syndromes of behavior problems. The Spanish YSR scales have shown good internal consistency (alpha > .90) in our past work with Hispanic adolescents. The YSR takes about 25 minutes to administer.
Change in Youth Outcome Questionnaire (YOQ) | At baseline and 4, 10, and 16 months post randomization.
  The Interpersonal Relations and Social Problems scales from the YOQ (Burlingame, Wells, & Lambert, 1996) will be used in this study. The YOQ was developed for children and adolescents ages 4-17 to track therapeutic progress. The Interpersonal Relations scale measures children's interactions, aggressiveness, and arguments with peers and adults. The Social Problems scale measures problematic behaviors such as running away, truancy, and destroying property. Internal consistency estimates of subscales range from .74 to .93 with a total scale score of .96.
Change in Parenting Practices Questionnaire (PPQ) | At baseline and 4, 10, and 16 months post randomization.
  The PPQ (Gorman-Smith et al., 1995) assesses four dimensions of parenting behavior: positive parenting, discipline effectiveness, discipline avoidance, and extent of involvement. Parents report on all four dimensions; adolescents report only on positive parenting and extent of involvement. The reliability of the PPQ has been supported by confirmatory factor analysis, with internal consistency coefficients ranging from .68 to .81. In our work with Hispanic adolescents, the PPQ subscales showed acceptable internal consistency (alpha) coefficients (.74 to .93).
Change in Parental Monitoring Instrument (PMI) | At baseline and 4, 10, and 16 months post randomization.
  The PMI (Cottrell et.al. 2007) was developed to determine how often parents use seven monitoring strategies: direct monitoring, indirect monitoring, school, health, computer, phone, and restrictive. The scale contains 27 items with 4 frequency responses (0 times, 1 to 2 times, 3 to 4 times, and 5-plus times). Parents and adolescents report how many times parents used a specific monitoring strategy in the past 4 months. In the development study, PMI has shown acceptable internal consistency (alpha) coefficients for parents (.71 to .85) and adolescents (.71 to .81).
Change in Family Environment Scale (FES) | At baseline and 4, 10, and 16 months post randomization.
  The FES is a brief 18-item self-report scale (Moos & Moos, 1994). Only two subscales are used in this study. The Cohesion scale measures the extent to which the adolescent or parent views the family as harmonious and close. The Conflict scale measures the extent to which the adolescent or parent views the family as characterized by frequent quarrels and disagreements. In our work with Hispanic adolescents, the FES showed acceptable internal consistency (alpha) coefficients (.69 to .81) and test-retest reliability (.85 to .86) at two-months.
Change in Inventory of Parent and Peer Attachment (IPPA) | At baseline and 4, 10, and 16 months post randomization.
  The IPPA (Armsden & Greenberg, 1987) is a self-report measure of adolescents' perception of their attachment to their parents along three dimensions: degree of mutual trust, quality of communication and the extent of anger and alienation. Internal consistency (alpha) coefficients are .87 for the mother version and .89 for the father version.
Change in Parent Barriers to Talk About Sex | At baseline and 4, 10, and 16 months post randomization.
  Parents will be administered 31 items from a larger measure used in the National Longitudinal Adolescent Health Questionnaire, which ask about parental attitudes and behaviors with regards to speaking with their adolescents about sex and birth control (Bearman, Jones, Jo, & Udry, 1997).
Change in Caregiver strain questionnaire (CGSQ) | At baseline and 4, 10, and 16 months post randomization.
  The CGSQ measures self-reported strain experienced by caregivers and families of youth. For each of the scale's 21 items, caregivers are asked to rate how much of a problem each item was for them. Impact areas covered by the CGSQ include family relations, time demands, psychological adjustment, financial burden, stigma, anger, and worry/guilt.
Change in Working Alliance Inventory (WAI) | At baseline and 4, 10, and 16 months post randomization.
  The WAI (Horvath and Greenberg, 1989) is a 10-minute measure of the quality and strength of the alliance between therapist and client on three dimensions: Goal, Task, and Bond. Reported reliabilities for the therapist version were .87 for the Goal scale, .82 for the Task scale and .68 for the Bond scale. For the client version, reliabilities of .89 for the Goal scale, .92 for both the Task and Bond scale.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A. Santisteban, Ph.D., Principal Investigator — University of Miami; Maite P. Mena, Psy.D., Study Director — University of Miami
Locations (1):
- Gables Waterway Executive Center (Clinic), Miami, Florida, United States

REFERENCES:
- [Background] Huey SJ Jr, Polo AJ. Evidence-based psychosocial treatments for ethnic minority youth. J Clin Child Adolesc Psychol. 2008 Jan;37(1):262-301. doi: 10.1080/15374410701820174. PMID 18444061
- [Background] Santisteban DA, Mena MP, McCabe BE. Preliminary results for an adaptive family treatment for drug abuse in Hispanic youth. J Fam Psychol. 2011 Aug;25(4):610-4. doi: 10.1037/a0024016. PMID 21639636
- [Background] Santisteban DA, Mena MP. Culturally informed and flexible family-based treatment for adolescents: a tailored and integrative treatment for Hispanic youth. Fam Process. 2009 Jun;48(2):253-68. doi: 10.1111/j.1545-5300.2009.01280.x. PMID 19579908
- [Background] Santisteban DA, Tejeda M, Dominicis C, Szapocznik J. An efficient tool for screening for maladaptive family functioning in adolescent drug abusers: the Problem Oriented Screening Instrument for Teenagers. Am J Drug Alcohol Abuse. 1999 May;25(2):197-206. doi: 10.1081/ada-100101855. PMID 10395155
- [Background] Santisteban, D., Szapocznik, J., Perez-Vidal, A., Kurtines, W. M., Coatsworth, J.D., et al. (1996). Efficacy of intervention for engaging youth and families into treatment and some variables that may contribute to differential effectiveness. Journal of Family Psychology, 10, 35-44.
- [Background] Santisteban, D.A., & Szapocznik, J. (1994). Bridging theory, research and practice to more successfully engage substance abusing youth and their families into therapy. Journal of Child and Adolescent Substance Abuse, 32 (2), 9-24.
- [Background] Szapocznik, J., Hervis, O., & Schwartz, S. (2003) Brief Stategic Family Therapy for Adolescent Drug Abuse. Therapy Manuals for Drug Addiction. U.S. Department of Health and Human Services. Bethesda, Maryland.
- [Background] Santisteban DA, Muir JA, Mena MP, Mitrani VB. INTEGRATIVE BORDERLINE ADOLESCENT FAMILY THERAPY: MEETING THE CHALLENGES OF TREATING ADOLESCENTS WITH BORDERLINE PERSONALITY DISORDER. Psychotherapy (Chic). 2003 Winter;40(4):251-264. doi: 10.1037/0033-3204.40.4.251. PMID 25663719
- [Background] Bry BH, Krinsley KE. Booster sessions and long-term effects of behavioral family therapy on adolescent substance use and school performance. J Behav Ther Exp Psychiatry. 1992 Sep;23(3):183-9. doi: 10.1016/0005-7916(92)90035-h. PMID 1487536